CLINICAL TRIAL: NCT06870045
Title: Investigation of Validity and Reliability of Dynamic Walking Index in Childhood Rheumatic Diseases
Brief Title: Dynamic Gait Index as a Functional Gait Assessment Measure in Children With JIA
Status: Recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Medipol University (Other); Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Gokce Leblebici, Assistant Professor, Istanbul University - Cerrahpasa
Other Study IDs: dyi_jia
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Juvenile Idiopathic Arthritis; Childhood Rheumatic Disease
Keywords: juvenile idiopathic arthritis; gait; dynamic gait index; childhood rheumatic diseases
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: This group will be created with children with juvenile idiopathic arthritis.
  Interventions: Other: Physical examination; Other: Dynamic Gait Index
- Healthy control group: This group will be created with age matched healthy volunteers.
  Interventions: Other: Dynamic Gait Index

INTERVENTIONS:
Other: Physical examination — The physical examination will included Timed Up and Go Test (TUG), Walking speed, Wong-Baker FACES Pain Scale, Pediatric balance scale and CHAQ (Childhood Health Assessment Questionnaire).
  Groups: Patient group
Other: Dynamic Gait Index — The DGI, whose validity and reliability will be investigated, consists of 8 items: walking on level ground, walking with changing speed, walking with sideways head turns, walking with vertical head turns, walking with pivot turns, walking over obstacles, going around obstacles, and climbing stairs. Performance on each item is rated on a 4-point scale ranging from 0 (severe impairment) to 3 (normal walking ability without a walking aid). The total score is 24. Scores below 19 indicate a risk of falling, while scores above 22 define safe ambulation.

SUMMARY:
Juvenile idiopathic arthritis (JIA) is one of the most common chronic rheumatic diseases seen in childhood. Pain, joint swelling and loss of function caused by inflammation significantly reduce the patients' quality of life and lead to muscle weakness, limited range of motion and gait disorders. Although there are various clinical assessment methods, there is no functional test in the current literature that evaluates walking in children with JIA.

The Dynamic Gait Index (DGI) is a functional walking scale that evaluates walking on level ground, walking while changing speed, walking with sideways head turns, walking with vertical head turns, walking with pivot turns, walking by jumping over obstacles, going around obstacles and climbing stairs. While the DGA is widely used in the clinical assessment of walking in older adults and other pediatric patient groups, it has not yet been investigated for the assessment of walking difficulties in children with JIA. This study aimed to determine whether the DYI is a usable tool for assessing walking in children with JIA.

ELIGIBILITY:
Inclusion Criteria:

* Study Group;
* Having a JIA diagnosis according to ILAR criteria between the ages of 8-16,
* Having unilateral knee joint involvement that will affect walking
* Being compatible, volunteer and cooperative in the study Control Group;

  1. Not having any neurological or orthopedic diagnosis
  2. Being between the ages of 8-16
  3. Being at a mental level that can understand the commands of the person performing the evaluation

Exclusion Criteria:

* Study Group;
* Having an additional neurological or orthopedic diagnosis accompanying JIA and affecting treatment results,
* Having lower extremity asymmetry or active lower extremity involvement other than the knee joint that will affect walking.

Control Group;

-Having any health problem that may affect the study

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Juvenile Idiopathic Arthritis
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dynamic Gait Index | Baseline and after 2 weeks from the baseline evaluation
  The DGI consists of 8 items: walking on level ground, walking with changing speed, walking with sideways head turns, walking with vertical head turns, walking with pivot turns, walking over obstacles, going around obstacles, and climbing stairs. Performance on each item is rated on a 4-point scale ranging from 0 (severe impairment) to 3 (normal ability to walk without a walking aid). The total score is 24. Scores below 19 indicate a risk of falling, while scores above 22 describe safe ambulation.
Walking speed | Baseline
  For the walking speed assessment, participants will be asked to walk along a 10-meter walkway at their preferred speed. Before the test, participants will be asked to walk 5 laps on the walkway and will be allowed to get used to the environment. During the walk, a video recording will be made in order to calculate the walking speed. For each participant, a video recording will be made with a camera fixed on a tripod placed laterally. During the walk, the participant's walking speed will be evaluated with the Kinovea 2D motion analysis program (Kinovea 0.8.15., GPLv2 license, 2019). Participants will be asked to walk 7 laps along the walkway, and the average data of these laps and the time taken to walk the 10-meter walkway in each lap will be recorded.
Timed Up and Go Test | Baseline
  The TUG test measures the time it takes for a person to get up from an arm-supported chair, walk 3 m, walk back to the chair, and sit down. The person walks at the preferred speed in their usual shoes with or without a walking aid. The tester remains with the participants at all times to ensure safety. Before starting the movement, the movement is demonstrated and explained to the child. The time it takes to get up from the chair and sit back in it is recorded. The test is repeated twice and the fastest score is recorded. Times less than 10 seconds are considered normal, while times greater than 14 seconds are recorded as a high risk of falling.
Wong-Baker FACES Pain Scale | Baseline
  The Wong-Baker FACES Pain Scale is a pain rating scale used to show children their pain intensity levels. On this scale, a person who feels happy indicates that they feel no pain (no pain), while a person who feels sad indicates that they feel a little or a lot of pain, Face 0 is very happy because they feel no pain. Face 10 visually represents severe pain that leads to crying. Participants will be asked to choose the face that best describes their pain from the scale before and after taping to assess pain.
Pediatric Balance Scale | Baseline
  To detect balance loss in children, the Pediatric Balance Scale, which is a modified version of the Berg balance scale and is used to assess functional balance skills in school-aged children, will be applied. The scale consists of 14 items, scored from 0 (lowest function) to 4 (highest function), with a maximum score of 56. The Pediatric Balance Scale is designed for use in school-aged children with mild to moderate motor impairments. Pilot testing was conducted on children aged 5 to 15 years.

SECONDARY OUTCOMES:
Childhood Health Assessment Questionnarie | Baseline
  The questionnaire consists of two different sections, the disability index and the discomfort index. The disability index consists of 8 parameters including dressing and personal care, standing up, eating, walking, hygiene, reaching out, holding and activities. All of these areas were assessed in 3 components. 1) How much difficulty they had in performing which daily functions 2) Whether they used special devices for daily functions 3) Whether they needed help from someone else in these activities were asked from each patient. There are 4 different possibilities for answers: 0 = no difficulty, 1 = with some difficulty, 2 = with great difficulty, 3 = unable. Discomfort was assessed by measuring pain with a 15 cm visual analog scale. The parents of the patients were asked to rate how much pain their child had in the past week and to give a score between 0 and 100. Similarly, they are asked to score between 0 and 100 on how much they have been affected by the disease since its onset

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ozdogan H, Ruperto N, Kasapcopur O, Bakkaloglu A, Arisoy N, Ozen S, Ugurlu U, Unsal E, Melikoglu M; Paediatric Rheumatology International Trials Organisation. The Turkish version of the Childhood Health Assessment Questionnaire (CHAQ) and the Child Health Questionnaire (CHQ). Clin Exp Rheumatol. 2001 Jul-Aug;19(4 Suppl 23):S158-62. PMID 11510322
- [Background] Franjoine MR, Gunther JS, Taylor MJ. Pediatric balance scale: a modified version of the berg balance scale for the school-age child with mild to moderate motor impairment. Pediatr Phys Ther. 2003 Summer;15(2):114-28. doi: 10.1097/01.PEP.0000068117.48023.18. PMID 17057441
- [Background] Balsalobre-Fernandez C, Tejero-Gonzalez CM, del Campo-Vecino J, Bavaresco N. The concurrent validity and reliability of a low-cost, high-speed camera-based method for measuring the flight time of vertical jumps. J Strength Cond Res. 2014 Feb;28(2):528-33. doi: 10.1519/JSC.0b013e318299a52e. PMID 23689339
- [Background] Garra G, Singer AJ, Taira BR, Chohan J, Cardoz H, Chisena E, Thode HC Jr. Validation of the Wong-Baker FACES Pain Rating Scale in pediatric emergency department patients. Acad Emerg Med. 2010 Jan;17(1):50-4. doi: 10.1111/j.1553-2712.2009.00620.x. Epub 2009 Dec 9. PMID 20003121
- [Background] Williams EN, Carroll SG, Reddihough DS, Phillips BA, Galea MP. Investigation of the timed 'up & go' test in children. Dev Med Child Neurol. 2005 Aug;47(8):518-24. doi: 10.1017/s0012162205001027. PMID 16108451
- [Background] Lubetzky-Vilnai A, Jirikowic TL, McCoy SW. Investigation of the Dynamic Gait Index in children: a pilot study. Pediatr Phys Ther. 2011 Fall;23(3):268-73. doi: 10.1097/PEP.0b013e318227cd82. PMID 21829122
- [Background] Shumway-Cook A, Baldwin M, Polissar NL, Gruber W. Predicting the probability for falls in community-dwelling older adults. Phys Ther. 1997 Aug;77(8):812-9. doi: 10.1093/ptj/77.8.812. PMID 9256869
- [Background] Jonsdottir J, Cattaneo D. Reliability and validity of the dynamic gait index in persons with chronic stroke. Arch Phys Med Rehabil. 2007 Nov;88(11):1410-5. doi: 10.1016/j.apmr.2007.08.109. PMID 17964880
- [Background] Hall CD, Herdman SJ. Reliability of clinical measures used to assess patients with peripheral vestibular disorders. J Neurol Phys Ther. 2006 Jun;30(2):74-81. doi: 10.1097/01.npt.0000282571.55673.ed. PMID 16796772
- [Background] Chiu YP, Fritz SL, Light KE, Velozo CA. Use of item response analysis to investigate measurement properties and clinical validity of data for the dynamic gait index. Phys Ther. 2006 Jun;86(6):778-87. PMID 16737403
- [Background] Herman T, Inbar-Borovsky N, Brozgol M, Giladi N, Hausdorff JM. The Dynamic Gait Index in healthy older adults: the role of stair climbing, fear of falling and gender. Gait Posture. 2009 Feb;29(2):237-41. doi: 10.1016/j.gaitpost.2008.08.013. Epub 2008 Oct 8. PMID 18845439
- [Background] Martini A. Systemic juvenile idiopathic arthritis. Autoimmun Rev. 2012 Nov;12(1):56-9. doi: 10.1016/j.autrev.2012.07.022. Epub 2012 Aug 2. PMID 22884552
- [Background] Ravelli A, Martini A. Juvenile idiopathic arthritis. Lancet. 2007 Mar 3;369(9563):767-778. doi: 10.1016/S0140-6736(07)60363-8. PMID 17336654
- [Background] Martini A, Lovell DJ, Albani S, Brunner HI, Hyrich KL, Thompson SD, Ruperto N. Juvenile idiopathic arthritis. Nat Rev Dis Primers. 2022 Jan 27;8(1):5. doi: 10.1038/s41572-021-00332-8. PMID 35087087